CLINICAL TRIAL: NCT06191588
Title: Feasibility and Effectiveness of Home-base Early Intensive Therapy in Unilateral Cerebral Palsy (Ucp-HEIT) Under-2-years-old
Brief Title: Intensive Therapies to Improve Manipulation in Young Children With Hemiparesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Elena Piñero Pinto, Professor, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USeville23
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Infantile Hemiplegia; Constraint Induced Movement Therapy; Family; Bimanual Intensive Therapy
MeSH Terms: conditions — Hemiplegia | interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- infant cimt (Experimental): Other: Infant BIT Not use of unaffected hand containment. Both hand are use to improve the bimanual coordination
  Other: Infant CIMT/BIT Use unaffected hand containment in part of the intervention and then, both hands in bimanual activities without containment.
  Other: Conventional therapy Following the usual therapy in the baby.
  Interventions: Procedure: INFANT CIMT/BIT
- Infant BIT (Active Comparator): Other: Infant CIMT/BIT Use unaffected hand containment in part of the intervention and then, both hands in bimanual activities without containment.
  Other: Conventional therapy Following the usual therapy in the baby.
  Other: infant cimt use of unaffected hand containment to improve the use of affected hand with unimanual activities
  Interventions: Procedure: INFANT CIMT/BIT
- Infant CIMT/BIT (Active Comparator): Other: Infant CIMT/BIT Use unaffected hand containment in part of the intervention and then, both hands in bimanual activities without containment.
  Other: Conventional therapy Following the usual therapy in the baby.
  Other: infant cimt use of unaffected hand containment to improve the use of affected hand with unimanual activities
  Interventions: Procedure: INFANT CIMT/BIT
- Conventional Therapy (Active Comparator): Other: Infant BIT Not use of unaffected hand containment. Both hand are use to improve the bimanual coordination
  Other: Infant CIMT/BIT Use unaffected hand containment in part of the intervention and then, both hands in bimanual activities without containment.
  Other: infant cimt use of unaffected hand containment to improve the use of affected hand with unimanual activities
  Interventions: Procedure: INFANT CIMT/BIT

INTERVENTIONS:
Procedure: INFANT CIMT/BIT — Constraint induced movement therapy (CIMT) and Bimanual Intensive therapy (BIT)
  Other Names: Constraint induced movement therapy; Bimanual Intentive Therapy

SUMMARY:
mCIMT and BIT are therapies applied in children with hemiplegia which have a great evidence, but not in a early age. This research has the objective to know the effects of this therapies in infants diagnosed of infantile hemiplegia from 9 to 18 months applying 50 hours of dose for both interventions during 10 weeks, executing them at home by families.

ELIGIBILITY:
Inclusion Criteria:

* Infantile hemiplegia
* Age from 9 months to 18 months.
* No use of the affected upper limb

Exclusion Criteria:

* Associated pathologies
* Epilepsy no controlled with drugs
* No collaborated families

Ages: 9 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
mini Assisting Hand Assesment | 10 weeks
  Bimanual functional performance Assessment in children with hemiplegia from 8 to 18 months.

SECONDARY OUTCOMES:
Satisfaction questionnaire for families | 10 weeks
  Descriptive questionnaire to obtain the adherence and satisfaction from families in this therapies.

CONTACTS AND LOCATIONS:
Locations (1):
- Elena Piñero Pinto, Seville, Spain

IPD SHARING:
Plan to Share IPD: Yes
Sharing data
Supporting Information: Study Protocol
Time Frame: For a year since the study ends

REFERENCES:
- [Derived] Palomo-Carrion R, Pinero-Pinto E, Lirio-Romero C, Romay-Barrero H, Ferri-Morales A, Romero-Galisteo RP. Home-based early intensive manual therapy in unilateral cerebral palsy under 2 years of age. Pediatr Res. 2025 Jul 26. doi: 10.1038/s41390-025-04306-4. Online ahead of print. PMID 40715358